CLINICAL TRIAL: NCT00053690
Title: Cognitive-Behavioral Treatment of PTSD in SMI Clients
Brief Title: Treatment of Post Traumatic Stress Disorder in Patients With Other Mental Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH064662-01 (NIH); R01MH064662-01 (NIH); DSIR AT-SP
Record Dates: First submitted 2003-02-04; First posted 2003-02-05 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2009-02

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Comorbidity; Schizophrenia; Bipolar Disorder; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Schizophrenia; Bipolar Disorder; Depression

INTERVENTIONS:
Behavioral: Cognitive Behavior Treatment

SUMMARY:
The purpose of this study is to develop an effective treatment for people with Post Traumatic Stress Disorder (PTSD) along with other mental illnesses.

DETAILED DESCRIPTION:
Despite the progress in treating PTSD in the general population and the elevated prevalence of PTSD in people with severe mental illness (SMI), there are no empirically validated treatments designed for patients with comorbid PTSD. The cognitive behavioral treatment provided in this study may improve knowledge of PTSD, decrease distorted beliefs, reduce PTSD symptoms, and improve quality of life.

Participants are randomly assigned to receive either a cognitive behavioral treatment plus standard care for SMI or standard care alone. The cognitive behavioral treatment incorporates several common features, including psychoeducation, relaxation training, and cognitive restructuring. Standard care for SMI includes medication, case management, and psychosocial treatment. PTSD, psychiatric symptoms, health, quality of life, and substance abuse outcomes are measured. Participants' knowledge of PTSD and beliefs about the world are also measured. Participants are assessed at baseline, post-treatment (16 weeks), and at 3- and 6-month follow-ups.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00494650

ELIGIBILITY:
Inclusion Criteria:

* Post Traumatic Stress Disorder
* New Hampshire definition of SMI plus DSM-IV Axis I diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depression
* Case management services and contact with a case manager at least twice a week

Exclusion Criteria:

* Alcohol or drug dependence
* Hospitalization or suicide attempt in the past 2 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88
Dates: Start 2002-01; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Kim Mueser, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center; Stanley Rosenberg, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Community Mental Health Centers in NH, Claremont, New Hampshire, United States

REFERENCES:
- [Derived] Mueser KT, McGurk SR, Xie H, Bolton EE, Jankowski MK, Lu W, Rosenberg SD, Wolfe R. Neuropsychological predictors of response to cognitive behavioral therapy for posttraumatic stress disorder in persons with severe mental illness. Psychiatry Res. 2018 Jan;259:110-116. doi: 10.1016/j.psychres.2017.10.016. Epub 2017 Oct 6. PMID 29040946